CLINICAL TRIAL: NCT05800275
Title: Multicentric Single Arm Phase II Study Evaluating the Efficacy of Association of Tucatinib, Capecitabine and Intra-CSF Trastuzumab in HER2 Amplified Breast Cancer Patients With Leptomeningeal Metastases
Brief Title: Capecitabine, Tucatinib, and Intrathecal Trastuzumab for Breast Cancer Patients With Leptomeningeal Disease
Acronym: ETIC-LM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-BCG-2205; 2022-001529-61 (EudraCT Number); 2022-502351-60-00 (Other: EU CT number)
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Leptomeningeal Metastasis; Leptomeningeal Disease; HER2-positive Metastatic Breast Cancer
Keywords: Intrathecal injection; Leptomeningeal Disease; Breast Cancer Metastatic; Leptomeningeal Metastasis; Intrathecal trastuzumab; Capecitabine; Tucatinib; HER2-positive Metastatic Breast Cancer
MeSH Terms: conditions — Meningeal Carcinomatosis; Meningeal Neoplasms | interventions — tucatinib; Capecitabine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tucatinib + Intrathecal Trastuzumab + Capecitabine (Experimental): Intra-CSF trastuzumab: 150 mg weekly Tucatinib: 300 mg orally twice daily Capecitabine: 1000 mg/m² orally twice daily on days 1-14 of each 21-day cycle
  Interventions: Drug: Tucatinib Oral Tablet; Drug: Capecitabine tablets; Drug: Trastuzumab Injection

INTERVENTIONS:
Drug: Tucatinib Oral Tablet — 300 mg, twice daily
Drug: Capecitabine tablets — 1000 mg/m², twice daily on days 1-14 of each 21-day cycle
Drug: Trastuzumab Injection — Intrathecal by lumbar puncture or Ommaya Reservoir, 150 mg weekly

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of tucatinib and capecitabine in combination with intrathecal trastuzumab on overall survival rate at 12 months in HER2-positive metastatic breast cancer (MBC) patients with proven leptomeningeal evolution and requiring intrathecal therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed a written informed consent form prior to any trial specific procedures. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent;
2. Patients ≥18 years old;
3. Histologically confirmed metastatic breast cancer;
4. Histologically confirmed HER2 positive breast cancer, with HER2 positive defined by in situ hybridization (ISH), immunohistochemistry (IHC), or fluorescence in situ hybridization (FISH) methodology; Note: HER2 testing should be performed preferably metastatic site; any estrogen and progesterone (ER/PR) status is allowed;
5. Proven leptomeningeal progression defined by linear leptomeningeal metastases on magnetic resonance imaging (MRI) or the presence of breast cancer cells in CSF (obtained within 28 days before inclusion );
6. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-2;
7. Life expectancy ≥2 months;
8. Stable dose of steroids for at least 5 days prior to registration;
9. If symptomatic brain or leptomeningeal metastasis, local treatment (surgery, radiation therapy) is allowed until 2 weeks before inclusion but should have been completed no more than 8 weeks before inclusion and with no clinical indication for immediate re-treatment with local therapy in the opinion of the investigator;
10. Adequate hematological function within 14 days before inclusion: Absolute neutrophil count (ANC) ≥1.5 x 10⁹/L; platelets count ≥100 x 10⁹/L; and hemoglobin ≥9.0 g/dL;
11. Adequate liver function within 14 days before inclusion: total bilirubin ≤1.5 ULN (unless documented Gilbert's syndrome); AST and ALT ≤2.5 ULN (≤5 ULN in the presence of liver metastases);
12. Normal renal function within 14 days before inclusion: estimated creatinine clearance ≥60 mL/min according to the Cockcroft-Gault formula;
13. Adequate cardiac function:

    * 12 Lead electrocardiograms (ECG) with normal tracing or non-clinically significant changes that do not require medical intervention
    * QT/QTc interval ≤470 msec for woman and ≤450 msec for men (mean of replicate values, correction per institutional standard) on the ECG at the screening visit and a normal kaliemia
    * Left ventricular ejection fraction (LVEF) ≥55%
    * No history of Torsades de Pointes or other symptomatic QTc abnormality
14. Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to National cancer institute-Common terminology criteria for adverse events (NCI-CTCAE) version 5.0 grade 1 or 0 to baseline (except alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion);
15. Women of childbearing potential must have a negative pregnancy test (blood or urine test) within 14 days prior to inclusion;
16. Woman of childbearing potential and male patients must agree to use adequate contraception for the duration of trial participation and up to 7 months after completing treatment/therapy. Hormonal contraceptives such as birth control pills, patches, implants, or injections are not allowed in patients who are hormone receptor positive;
17. Patients affiliated to the social security system (or equivalent);
18. Patient must be willing and able to comply with the protocol for the duration of the trial including scheduled visits, treatment plan, laboratory tests, and examinations including follow-up.

Exclusion Criteria:

1. Used of a strong cytochrome P450 (CYP)2C8 inhibitor within 5 half-lives of the inhibitor, or use of a strong CYP3A4 or CYP2C8 inducer within 5 days prior to first dose of study treatment. Use of sensitive CYP3A substrates should be avoided one week before enrollment and during study treatment;
2. Previous treatment with Tucatinib or Capecitabine;
3. Severe leukopenia, neutropenia, or thrombocytopena, severe hepatic impairment, severe renal impairment (creatinine clearance below 30mL/min)
4. Recent or concomitant treatment with brivudine ;
5. Any antiplatelet or curative anticoagulant treatment for blood coagulation disorders;
6. Severe pre-existing cerebrovascular dysfunction or pathology such as stroke and intra-cerebral hematoma or uncontrolled intracerebral hypertension induced by brain metastasis;
7. Ventriculoperitoneal or atrial shunt, except if the valve is equipped with an on-off device and that the patient's condition allows for to remain in the off position for 6 hours after each injection of trastuzumab;
8. Known history of testing positive for HIV or known acquired immunodeficiency syndrome;
9. Carriers of Hepatitis B or Hepatitis C or have other known chronic liver disease;
10. Uncontrolled hypertension;
11. Uncontrolled infection;
12. Severe dyspnea at rest due to complications of advanced malignancy or requiring supplementary oxygen therapy;
13. Pregnant or breast-feeding women;
14. Known prior severe hypersensitivity to tucatinib or compounds chemically or/and biologically similar or any component in its formulation;
15. Hypersensitivity to trastuzumab, murine proteins, or to any of the excipients in its formulation;
16. Known prior severe hypersensitivity to capecitabine or to any of the excipients or fluorouracil;
17. Known complete dihydropyrimidine dehydrogenase (DPD) deficiency (if applicable);
18. Inability to swallow tablets or significant gastrointestinal disease which would preclude the adequate oral absorption of medications;
19. Prior history of other malignancies other than study disease (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) unless the patient has been free of the disease for at least 5 years;
20. Person deprived of their liberty or under protective custody or guardianship;
21. Participation in another therapeutic trial within the 30 days prior to treatment initiation;
22. Patients with any other disease or illness, which requires hospitalization or is incompatible with the trial treatment, are not eligible. Patients unwilling or unable to comply with trial obligations for geographic, social, or physical reasons, or who are unable to understand the purpose and procedures of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
overall survival rate at 12 months | 12 months
  12-month overall survival will be defined as the proportion of patients alive 12 months after treatment initiation.

SECONDARY OUTCOMES:
Clinical neurological symptoms relief | At baseline, every week during treatment up to 18 months then every 9 weeks up to 42 months
  Clinical neurological symptoms relief will be defined as complete or partial diminution of symptoms associated to leptomeningeal metastasis using the neurologic assessment in neuro-oncology (NANO) scale, a standardized questionnaire designed to measure neurological function in oncology.
  The questionnaire includes 5 domains scored 0-3 (gait, strength, visual fields, language, and level of consciousness) and 4 domains scored 0-2 (ataxia of upper extremities, sensation, facial strength, and behavior). Scores are sum up to a maximum of 23 points with high-scale values representing impaired neurological performances.
Progression free survival (PFS) | From inclusion to disease progression or death, up to 42 months
  The progression-free survival (PFS) is the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse.
Overall survival (OS) | From inclusion to death from any cause; up to 42 months
  The overall survival (OS) is the length of time from inclusion in the study that patients are still alive.
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline, every 3 weeks during treatment up to 18 months then every 9 weeks up to 42 months
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life Questionnaire - Brain Cancer Module (QLQ-BN20) | At baseline, every 3 weeks during treatment up to 18 months then every 9 weeks up to 42 months
  This EORTC brain cancer specific questionnaire is intended to supplement the QLQ-C30.
  The QLQ-BN20 contains 20 items organized into four scales (three items each: future uncertainty, visual disorder, motor dysfunction, and communication deficit), and seven single items (headaches, seizures, drowsiness, hair loss, itchy skin, weakness of legs, and bladder control). All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale, with higher scores indicating more severe symptoms.
Intra-cerebrospinal fluid response at 4 weeks | 4 weeks
  Intra-cerebrospinal fluid (CSF) response at 4 weeks will be defined by absence, evaluated by the cytologist, of tumor cells in the intra-cerebrospinal fluid of the patient.
Duration of leptomeningeal metastases (LM) response | From inclusion to disease LM progression or death, up to 42 months
  Duration of LM response is the length of time from first intracranial objective response and disease progression.
  For this outcome, disease progression is defined as the length of time during and after the treatment of a disease that a patient lives with the leptomeningeal metastases but they does not get worse.
Montreal Cognitive Assessment (MoCA) | At baseline, every 3 weeks during treatment up to 18 months then every 9 weeks up to 42 months
  The Montreal Cognitive Assessment (MoCA) is a widely used screening assessment for detecting cognitive dysfunctions.
  The test is a 30-point test assesses different cognitive domains: attention and concentration (5 points), executive functions (4 points), memory (2 points), language (5 points), visuospatial skills (4 points), conceptual thinking (1 point), calculations (3 points), and orientation (6 points). MoCA scores range between 0 and 30, a score of 26 or over is considered normal.
Toxicity during the study | Throughout study completion, up to 42 months
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Louis LARROUQUERE, Principal Investigator — Centre Léon Bérard, Lyon
Locations (11):
- France (11):
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges-François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Institut régional du Cancer de Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Institut de cancérologie Strasbourg Europe - ICANS, Strasbourg
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.